CLINICAL TRIAL: NCT04716868
Title: Prospective, Randomized and Controlled Study for the Evaluation of the Effectiveness of a Supplement of Agave Tequilana Weber Var. Azul Fiber Derivatives vs Psyllium Plantago in Patients With Functional Constipation
Brief Title: Evaluation of a Supplement of Agave Tequilana Weber Azul vs Psyllium Plantago in Patients With Functional Constipation
Acronym: SATWAVPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Enrique Coss-Adame, Gastroenterology, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAS-1107-13/15-1
Record Dates: First submitted 2019-10-17; First posted 2021-01-20 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Functional Constipation
Keywords: Functional constipation; Agave tequilana Weber var. Azul; Psyllium plantago; Microbiota
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: a prospective, randomized, controlled and single blind study to determine the efficacy of the blue agave Tequilana Weber fructans intake in subjects with functional constipation.
Who Masked: Participant, Investigator
Masking Description: Powder is flavored in order to mask at minimum the differences between type of fibers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Agave Fructans 5 g (Experimental): Agave tequilana Weber blue variety 5 g once a day for 8 week.
  Interventions: Dietary Supplement: Agave Fructans 5 g
- Agave Fructans 10 g (Experimental): Agave tequilana Weber blue variety 10 gf once a day for 8 week.
  Interventions: Dietary Supplement: Agave Fructans 10 g
- Maltodextrin 10 g + Agave Fructans 5 g (Experimental): Maltodextrin 10 g + Agave tequilana Weber blue variety 5 g once a day for 8 week.
  Interventions: Dietary Supplement: Agave Fructans 5 g + Maltodextrin 10 g
- Psyllium plantago 15 g (Active Comparator): Psyllium plantago 15 g once a day for 8 week.
  Interventions: Dietary Supplement: Psyllium plantago

INTERVENTIONS:
Dietary Supplement: Agave Fructans 5 g — Agave tequilana Weber blue variety 5 g once a day for 8 weeks
  Other Names: Agave fructans
  Arms: Agave Fructans 5 g
Dietary Supplement: Agave Fructans 10 g — Agave tequilana Weber blue variety 10 g once a day for 8 weeks
  Other Names: Agave fructans
  Arms: Agave Fructans 10 g
Dietary Supplement: Agave Fructans 5 g + Maltodextrin 10 g — Maltodextrin 10 g + Agave tequilana Weber blue variety 5 g once a day for 8 weeks
  Other Names: Agave fructans
  Arms: Maltodextrin 10 g + Agave Fructans 5 g
Dietary Supplement: Psyllium plantago — Psyllium plantago 15 g once a day for 8 weeks
  Arms: Psyllium plantago 15 g

SUMMARY:
Introduction: Constipation is one of the gastrointestinal disorders MOST frequent That Affects around 20% of the western population, being more frequent in the female gender (M1.5: H1). Constipation can be primary, When causes constipation associated With (medication, mechanical obstruction, spinal cord injury, etc.) and secondary. There are multiple therapeutic options for the management of constipation, changes in lifestyle Including, the intake of fiber, laxatives and pharmacological treatment and in selected cases (colonic inertia) surgery. The first option in the therapeutic management for Patients With constipation are changes in lifestyle, Among Which is the type of diet (increase in fiber intake, Which Has Been Associated With an improvement in the fecal matter and the evacuation frequency), liquid intake and exercise. Aim: To Evaluate the efficacy of the blue agave fructans Tequilana Weber in Patients With functional constipation Methods: This is a prospective, randomized, controlled and single blind study to determine the phase III efficacy of the blue agave fructans Tequilana Weber intake in subjects with functional constipation. In order to Achieve so, it is planned to include over 18 years of Patients age Fulfill the WHO as well as inclusion criteria The Rome III criteria for functional constipation. Statistical analysis plan: The data obtained will be analyzed with SPSS version 24. For continuous variables the results are presented in mean ± standard deviation when the variables are normally distributed or medians and percentiles otherwise and as frequency and percentages when they were categorical. For basal and subsequent comparison to the intra intervention groups, Student's t-test for paired samples (variables with normal distribution) or the Mann-Whitney U (variables without normal distribution) is used in the case of continuous variables and X2 or the McNemar test in the case of categorical variables. For comparison between groups ANOVA (variables with normal distribution) or Kruskal-Wallis (non-normal distribution variables) used for continuous variables and the same percentage of change obtained when the variables are continuous. Also an analysis of covariance (ANCOVA) was performed to control variables that might have an effect on the response variables.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled and single blind study to determine the phase III efficacy of the blue agave fructans Tequilana Weber intake in subjects with functional constipation.

In order to Achieve so, it is planned to include over 18 years of Patients age Fulfill the WHO as well as inclusion criteria The Rome III criteria for functional constipation. (See table below).

The phase of our study is designated based on article 66 of chapter II "On Pharmacological Research" of the Regulation of the General Law on Health in Research That defines PHASE III studies Follows as: It is the administration of a research drug to large groups of Patients (Usually external), to define ITS therapeutic utility and identification identify adverse reactions, interactions and external factors That May alter the pharmacological effect.

Patients of the institute will be called after invitations to Participate in Placing a protocol for Patients With constipation. Patients Who Have Not Been registered and meet the inclusion criteria May Also Participate.

The study to be Carried out will be Explained and read and, where appropriate', the informed consent will be signed by the Patient During the initial visit (Visit 1) of eligibility, Where the subject will be Given 2 questionnaires (see annexes), one They meet to determine if the ROME III criteria for functional constipation (FC) and another to ASSESS if the patient does not meet the criteria for irritable ROME III bowel syndrome (IBS) and a baseline breath test will be performed.

In Addition, the previous use of fiber supplements and laxatives, which must be suspended at Least 2 months prior to randomization, will be EVALUATED.

The subject will return to a second visit (Visit 2) (Which will depend on Whether the patient is taking laxatives or fiber supplements) for a complete physical evaluation and the fiber intake diary will be Assessed to determine the amount of fiber intake in the diet as well as the diary of evacuations and the SmartPill © will be Given and That way, the patient will return to the hospital to register the data after the capsule Having evacuated.

The patient will return a week later (Visit 3) on a 12 hour fast, the fiber intake and the evacuation diaries will be re-EVALUATED and will be EVALUATED They again by a nutritionist. A new breath test will be Carried out. The subject will be Asked to complete the SF-36 Quality of Life Questionnaire. A stool sample will be Collected for ITS analysis in Addition to a blood sample for determination of fasting glucose, glycosylated hemoglobin A1c, Insulin and full lipid profile.

The subjects will be randomized to receive one of four treatments That can be Psyllium plantago 15g, blue agave Tequilana Weber fructans at doses of 5, 10g and blue agave Tequilana Weber fructans at a dose of 5 g + 10 g excipient for a concentration of 33 % of blue agave fructans Tequilana Weber.

The randomization will be computer-generated with a participation number and the assignment of the treatment will be consecutive.

The product will be supplied in identical bottles With the same amount of powder in a container That will only be identifiable With the name of the protocol as well as the patient's number.

The patient will be provided with a measuring spoon to administer the amount of product Necessary for each of the doses (5, 10 and 15g respectively) or with envelopes Containing the exact Amounts Weighed.

The patient will be instructed to keep a diary of the diet, of the evacuations and a sheet to ASSESS adverse effects. The subject will return (Visit 4) at the end of a month ± 5 days on a 12 hour fast and Their adherence will be Assessed by product weight in the container subtracting the number of grams required daily ACCORDING TO the assignment of treatment.

The fiber intake diaries will be EVALUATED again by the nutritionist, the evacuation will Also be EVALUATED diary. A medical evaluation will be Carried out That includes questioning and physical evaluation. Subsequently, a blood sample will be to determine fasting glucose Obtained, glycosylated hemoglobin A1c, insulin and lipid profile and a full sample of excrement will be Obtained and SmartPill® will be Given.

The patient will Continue with the supplement in the same container and will be scheduled for a month later. In the end-of-treatment visit visit (visit 5), the fiber will be EVALUATED journals consumption again by a nutritionist and the evacuation will be EVALUATED diary as well.

A medical evaluation will be Carried out That includes questioning and physical evaluation and Their adherence will be Assessed by weighing the product in the container, subtracting the number of grams That it requires daily ACCORDING to the treatment assignment or delivery by the patient of the empty envelopes used.

Subsequently, a blood sample will be to determine fasting glucose Obtained, glycosylated hemoglobin A1c, insulin and lipid profile and a full sample will be Collected stool and breath test at the end will be Carried out.

For end of the visit, Which Will Be Carried out one month after stopping the treatment, the evacuation will be EVALUATED diary and a stool sample will be Collected and with it the intervention in the part of the study will end. Total The follow-up duration for each patient will be 3 months, enough time to observe and compare the effect of the fibers to be used. It is Important to mention That in recent studies Carried out by the same team and with blue agave Tequilana Weber fructans, effects on intestinal transit Have Been observed from the first week of intake, in fact this is one of the Reasons to focus the study on functional constipation and intestinal transit.

Breath test:

A breath test will be Carried out in order to measure hydrogen and methane Concentrations previously Exhaled In Patients randomized in visits 1 and 5.

In order to carry out the breath test gas chromatography equipment will be used, brand Quintron® Breath-tracker.

For That, The Patients will be Asked:

* Not to take antibiotics prior weeks At least to the test.
* Stop the intake of food rich in fibers and starches 24 h before the test.
* Not to take alcohol, or smoke
* Have a minimum of 8 hours fasting
* Perform oral hygiene before starting the test and during the performance of measurements.

This test lasts 3 hours, during which the patient can not leave the laboratory facilities motility, can not speak too much or sleep. Exhaled air samples are taken every 15 minutes during this period.

SmartPill®:

SmartPill® test will be conducted on visits 2 and 4.

Colonoscopy:

Is a tool which will be subject to scrutiny patients ≥55 years with newly diagnosed constipation or those where changes in bowel habits observed in this age group. This fundamental objective, rule out potentially serious diseases and not to delay the diagnosis of these during the research study. one colonoscopic study all patients who have constipation and any of the following characteristics will be used:

1. Diagnosis of constipation less than 1 year
2. Subjects ≥55 years who do not have colonoscopic evaluation in the last 3 years prior to study entry
3. Chronic but with alarm data (: Unexplained weight loss, recent transrectal bleeding <6 months, recent changes in the defecation pattern example) Constipation

Patients include:

Studies with fiber supplements (Psyllium, Plums8) Have included 25 to 30 patients per group to find differences between groups.

In total it is planned to include 60 patients randomized as follows: 15 patients receive fructans blue agave Tequilana Weber dose of 5 g, 15 patients received the dose of 10 g, 15 patients received the dose of 5g of agave fructans blue Tequilana Weber + 10 g excipient and 15 patients received 15 g plantago psyllium.

Gas Chromatography: (determination of short-chain fatty acid AGCC)

AGCC for determining ion detector flame will be used. The following steps are performed:

1. 50 uL ethyl butyrate is added to 1 g of faeces
2. 1 mL of hydrochloric acid was be added.
3. It is centrifuged at 3000 g for 10 minutes. The supernatant was removed.
4. Subsequently it is added 300 uL N-Methyl dibutil sililtrifluoroacetamide (MTBSTFA).
5. solution at 80 ° C for 20 min heat up.
6. It left undisturbed at room temperature for 24 hrs to ensure complete derivatization of lactic acid.
7. analyzing samples by gas chromatography according to method developed for specific samples will be performed.

Extraction of DNA from faeces, PCR amplification and bacterial 16S rRNA sequencing:

RRNA sequencing is the method of choice to determine high taxonomic relationships (gender up level). Because the 16S rRNA molecule contains highly variable regions, it is usually possible to find regions 20 to 30 bases that are completely unique to a single species of bacteria.

To perform the analysis, will collect in fecal specimens are sterile plastic containers. Immediately after collection, the samples will be transported to the laboratory in ice bucket 2 to 8 and then frozen at -73 ° C until processing.

DNA extraction was carried out following the instructions of the automated method NucliSENS® easyMAG® (BioMerieux, Durham, NC, USA) with a brief initial modification before automated process. Is weighed and suspended 200 mg of fecal matter of each sample in 0.3 mL of phosphate buffered saline solution-(8 mM Na2HPO4, 137 mM NaCl, 2.7 mM KCl, 1.5 mM KH2PO4 and) vigorous agitation for 30 seconds. 100 .mu.l of the suspension was placed in boiling 15 min and immediately frozen at 0 ° C on ice. Bacterial homogenate was centrifuged at 13,000 g for 10 min and the supernatant will be collected in tubes 500 .mu.l.

This specimen will be used for the isolation of DNA on automated equipment. PCR amplification real time 16S rRNA bacterial be carried out as described by previous reports using a Light Cycler-(Roche) equipment.

Quantification of bacterial phyla in major categories described: 1) Firmicutes, 2) Bacteroidetes, 3) Actinobacterias, 4) Proteobacteria. It will be conducted by the method of quantitative PCR in real time using the primers and conditions described previously, pR amplify specific fragments of bacterial 16S rRNA population groups described. We will use primers called barcode 967 F (CNACGCGAAGAACCTTANC) and 1046R (CGACAGCCATGCANCACCT) to amplify the 16S rRNA fragments V6 bacterial V6.

Sequencing and analysis of the amplified fragments is by fluorescent sequencing equipment terminator 3130 / genetic analyzer (Applied Biosystems).

The PCR products were sequenced and analyzed and will be submitted to GenBank for species identification.

Extracting bacterial DNA and quantitation of bacterial species used to demonstrate the prebiotic effect of agave fiber, since selective growth of the population of bifidobacteria and lactobacilli and occurrence of short-chain fatty acid in stool is expected.

Thus in addition to the functional properties and their effects on constipation, you may check the prebiotic effect of agave fructans.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* functional constipation ROME III criteria as
* Subjects ≥55 years with recent colonoscopy (<3 years)

Exclusion Criteria:

* Taking supplements of fiber in the last 2 months
* Stimulant laxatives consumption chronically (Senna, Bisacodyl)
* decompensated comorbidities (example: uncontrolled diabetes mellitus HbA1c> 9%, decompensated Organ failure, decompensated hypertension (untreated or TA> 160 mmHg systolic and 95 mmHg diastolic)
* Using digital maneuvers or enemas to achieve evacuation
* Personal history of active or previous cancer
* abdominal surgery (except appendectomy, cholecystectomy, hysterectomy)
* Presence of alarm data in the last 6 months (trans-rectal bleeding, unexplained weight loss, abdominal pain)
* Use of drugs known promote constipation (opioid derivatives, calcium channel blockers, anticholinergics tricyclic antidepressants type)
* Prostration (immobility or poor mobility)
* Diseases such as untreated hypothyroidism with hormone replacement, and diseases associated with hypercalcemia that promote constipation
* Other causes of secondary constipation
* Meet criteria for constipation predominant irritable bowel
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2021-06-18 (Estimated); Study Completion 2021-08-18 (Estimated)

PRIMARY OUTCOMES:
An increase of more than one complete evacuation from basal spontaneous from baseline at the end of active | 15 days
  Effect of supplementation of fructans Tequilana Weber blue agave in increasing at least one complete evacuation from basal spontaneous. Spontaneous evacuation It is defined as an evacuation in the absence of use of laxatives, suppositories or enemas and complete evacuation is defined as spontaneous evacuation to that sensation of incomplete emptying of the rectal ampulla.

SECONDARY OUTCOMES:
Change in the classification of Bristol | 15 days
  Effect of supplementation of fructan Weber blue agave Tequilana in the form of bowel movements, assessed by the Bristol scale. It is defined as a change in the form of evacuations when presenting a change in the classification of Bristol, more than 50% according to the daily evacuations taking the average of the evacuations submitted within 15 days.
Effect of supplementation of fructan Weber blue agave Tequilana in the frequency of bowel movements | 15 days
  II. Effect of supplementation of fructan Weber blue agave Tequilana in the frequency of bowel movements. It shall be defined as responder presenting increased 50% in stool frequency compared with baseline, according to the daily bowel movements taking the average of evacuations presented at 15 days.
Evaluate the impact of the concentration of short-chain fatty acid, particularly butyrate, in the feces of subjects before and after addition of fructans Tequilana Weber blue agave. | 8 weeks
  The butyrate concentration was determined by method of gas chromatography and the increase will be assessed in millimoles per liter.
IV. Evaluate the impact of supplementation fructans Weber blue agave Tequilana the microbiota | 8 weeks
  determining edges present in feces of the subjects before and after the supplementation fructan derivatives fiber; which are: actinobacteria, bacteroidetes, firmicutes, proteobacteria and euryarchaeota
V. To evaluate the impact of serum glucose concentration and HbA1c fasting serum of subjects before and after addition of fructans Tequilana Weber blue agave | 8 weeks
  HbA1c concentration is determined as it is intended to monitor the impact of fiber on glucose throughout the duration of the study (2 months) and in order to avoid the variability that fasting glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Coss-Adame, Principal Investigator — National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Locations (1):
- National Institute of Medical Sciences and Nutrition Salvador Zubiran, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Remes Troche JM, Remes Troche JM, Tamayo de la Cuesta JL, Rana Garibay R, Huerta Iga F, Suarez Moran E, Schmulson M; Asociacion Mexicana de Gastroenterologia. [Guidelines for diagnosis and treatment of constipation in Mexico. A) Epidemiology (meta-analysis of the prevalence), pathophysiology and classification]. Rev Gastroenterol Mex. 2011 Apr-Jun;76(2):126-32. Spanish. PMID 21724488
- [Result] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Result] American Gastroenterological Association; Bharucha AE, Dorn SD, Lembo A, Pressman A. American Gastroenterological Association medical position statement on constipation. Gastroenterology. 2013 Jan;144(1):211-7. doi: 10.1053/j.gastro.2012.10.029. No abstract available. PMID 23261064
- [Result] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Result] Lopez-Colombo A, Morgan D, Bravo-Gonzalez D, Montiel-Jarquin A, Mendez-Martinez S, Schmulson M. The epidemiology of functional gastrointestinal disorders in Mexico: a population-based study. Gastroenterol Res Pract. 2012;2012:606174. doi: 10.1155/2012/606174. Epub 2012 Mar 19. PMID 22474443
- [Result] Eswaran S, Muir J, Chey WD. Fiber and functional gastrointestinal disorders. Am J Gastroenterol. 2013 May;108(5):718-27. doi: 10.1038/ajg.2013.63. Epub 2013 Apr 2. PMID 23545709
- [Result] Pucciani F, Raggioli M, Ringressi MN. Usefulness of psyllium in rehabilitation of obstructed defecation. Tech Coloproctol. 2011 Dec;15(4):377-83. doi: 10.1007/s10151-011-0722-4. Epub 2011 Jul 22. PMID 21779973
- [Result] Singh B. Psyllium as therapeutic and drug delivery agent. Int J Pharm. 2007 Apr 4;334(1-2):1-14. doi: 10.1016/j.ijpharm.2007.01.028. Epub 2007 Jan 21. PMID 17329047
- [Result] Xing JH, Soffer EE. Adverse effects of laxatives. Dis Colon Rectum. 2001 Aug;44(8):1201-9. doi: 10.1007/BF02234645. PMID 11535863
- [Result] Lopez MG, Mancilla-Margalli NA, Mendoza-Diaz G. Molecular structures of fructans from Agave tequilana Weber var. azul. J Agric Food Chem. 2003 Dec 31;51(27):7835-40. doi: 10.1021/jf030383v. PMID 14690361
- [Result] Urias-Silvas JE, Cani PD, Delmee E, Neyrinck A, Lopez MG, Delzenne NM. Physiological effects of dietary fructans extracted from Agave tequilana Gto. and Dasylirion spp. Br J Nutr. 2008 Feb;99(2):254-61. doi: 10.1017/S0007114507795338. Epub 2007 Aug 22. PMID 17711612
- [Result] Mellado-Mojica E, Lopez MG. Fructan metabolism in A. tequilana Weber Blue variety along its developmental cycle in the field. J Agric Food Chem. 2012 Nov 28;60(47):11704-13. doi: 10.1021/jf303332n. Epub 2012 Nov 14. PMID 23072425
- [Result] Guarner F. Enteric flora in health and disease. Digestion. 2006;73 Suppl 1:5-12. doi: 10.1159/000089775. Epub 2006 Feb 8. PMID 16498248
- [Result] Gerritsen J, Smidt H, Rijkers GT, de Vos WM. Intestinal microbiota in human health and disease: the impact of probiotics. Genes Nutr. 2011 Aug;6(3):209-40. doi: 10.1007/s12263-011-0229-7. Epub 2011 May 27. PMID 21617937
- [Result] Narvaez-Zapata JA, Sanchez-Teyer LF. Agaves as a raw material: recent technologies and applications. Recent Pat Biotechnol. 2009;3(3):185-91. doi: 10.2174/187220809789389144. PMID 19747148
- [Result] Escudero Alvarez E, Gonzalez Sanchez P. Dietary fibre. Nutr Hosp. 2006 May;21 Suppl 2:60-71, 61-72. English, Spanish. PMID 16771074
- [Result] Chierici R, Fanaro S, Saccomandi D, Vigi V. Advances in the modulation of the microbial ecology of the gut in early infancy. Acta Paediatr Suppl. 2003 Sep;91(441):56-63. doi: 10.1111/j.1651-2227.2003.tb00647.x. PMID 14599043
- [Result] Guarner F, Malagelada JR. Gut flora in health and disease. Lancet. 2003 Feb 8;361(9356):512-9. doi: 10.1016/S0140-6736(03)12489-0. PMID 12583961
- [Result] Tuohy KM, Rouzaud GC, Bruck WM, Gibson GR. Modulation of the human gut microflora towards improved health using prebiotics--assessment of efficacy. Curr Pharm Des. 2005;11(1):75-90. doi: 10.2174/1381612053382331. PMID 15638753
- [Result] Wang X, Gibson GR. Effects of the in vitro fermentation of oligofructose and inulin by bacteria growing in the human large intestine. J Appl Bacteriol. 1993 Oct;75(4):373-80. doi: 10.1111/j.1365-2672.1993.tb02790.x. PMID 8226394
- [Result] Kolida S, Tuohy K, Gibson GR. Prebiotic effects of inulin and oligofructose. Br J Nutr. 2002 May;87 Suppl 2:S193-7. doi: 10.1079/BJNBJN/2002537. PMID 12088518
- [Result] Schneeman BO. Fiber, inulin and oligofructose: similarities and differences. J Nutr. 1999 Jul;129(7 Suppl):1424S-7S. doi: 10.1093/jn/129.7.1424S. PMID 10395611
- [Result] Coussement PA. Inulin and oligofructose: safe intakes and legal status. J Nutr. 1999 Jul;129(7 Suppl):1412S-7S. doi: 10.1093/jn/129.7.1412S. PMID 10395609
- [Result] Carabin IG, Flamm WG. Evaluation of safety of inulin and oligofructose as dietary fiber. Regul Toxicol Pharmacol. 1999 Dec;30(3):268-82. doi: 10.1006/rtph.1999.1349. PMID 10620476
- [Result] Livesey G. Tolerance of low-digestible carbohydrates: a general view. Br J Nutr. 2001 Mar;85 Suppl 1:S7-16. doi: 10.1079/bjn2000257. PMID 11321031
- [Result] Bruhwyler J, Carreer F, Demanet E, Jacobs H. Digestive tolerance of inulin-type fructans: a double-blind, placebo-controlled, cross-over, dose-ranging, randomized study in healthy volunteers. Int J Food Sci Nutr. 2009 Mar;60(2):165-75. doi: 10.1080/09637480701625697. PMID 18608562
- [Result] Holscher HD, Doligale JL, Bauer LL, Gourineni V, Pelkman CL, Fahey GC, Swanson KS. Gastrointestinal tolerance and utilization of agave inulin by healthy adults. Food Funct. 2014 Jun;5(6):1142-9. doi: 10.1039/c3fo60666j. Epub 2014 Mar 25. PMID 24664349
- [Result] Marteau P, Flourie B. Tolerance to low-digestible carbohydrates: symptomatology and methods. Br J Nutr. 2001 Mar;85 Suppl 1:S17-21. doi: 10.1079/bjn2000258. PMID 11321024
- [Result] Avallone EV, De Carolis A, Loizos P, Corrado C, Vernia P. Hydrogen breath test--diet and basal H2 excretion: a technical note. Digestion. 2010;82(1):39-41. doi: 10.1159/000277630. Epub 2010 Feb 27. PMID 20197661
- [Result] Schneider AR, Jepp K, Murczynski L, Biniek U, Stein J. The inulin hydrogen breath test accurately reflects orocaecal transit time. Eur J Clin Invest. 2007 Oct;37(10):802-7. doi: 10.1111/j.1365-2362.2007.01862.x. Epub 2007 Aug 28. PMID 17727672
- [Result] Vilagut G, Ferrer M, Rajmil L, Rebollo P, Permanyer-Miralda G, Quintana JM, Santed R, Valderas JM, Ribera A, Domingo-Salvany A, Alonso J. [The Spanish version of the Short Form 36 Health Survey: a decade of experience and new developments]. Gac Sanit. 2005 Mar-Apr;19(2):135-50. doi: 10.1157/13074369. Spanish. PMID 15860162
- [Result] Chang L. Review article: epidemiology and quality of life in functional gastrointestinal disorders. Aliment Pharmacol Ther. 2004 Nov;20 Suppl 7:31-9. doi: 10.1111/j.1365-2036.2004.02183.x. PMID 15521853
- [Result] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Result] Bonnema AL, Kolberg LW, Thomas W, Slavin JL. Gastrointestinal tolerance of chicory inulin products. J Am Diet Assoc. 2010 Jun;110(6):865-8. doi: 10.1016/j.jada.2010.03.025. PMID 20497775
- [Result] Gomez E, Tuohy KM, Gibson GR, Klinder A, Costabile A. In vitro evaluation of the fermentation properties and potential prebiotic activity of Agave fructans. J Appl Microbiol. 2010 Jun;108(6):2114-21. doi: 10.1111/j.1365-2672.2009.04617.x. Epub 2009 Nov 4. PMID 19941629
- [Result] Holscher HD, Bauer LL, Gourineni V, Pelkman CL, Fahey GC Jr, Swanson KS. Agave Inulin Supplementation Affects the Fecal Microbiota of Healthy Adults Participating in a Randomized, Double-Blind, Placebo-Controlled, Crossover Trial. J Nutr. 2015 Sep;145(9):2025-32. doi: 10.3945/jn.115.217331. Epub 2015 Jul 22. PMID 26203099
- [Result] Ramnani P, Costabile A, Bustillo AG, Gibson GR. A randomised, double- blind, cross-over study investigating the prebiotic effect of agave fructans in healthy human subjects. J Nutr Sci. 2015 Mar 13;4:e10. doi: 10.1017/jns.2014.68. eCollection 2015. PMID 26090092
- [Result] Erdogan A, Rao SS, Thiruvaiyaru D, Lee YY, Coss Adame E, Valestin J, O'Banion M. Randomised clinical trial: mixed soluble/insoluble fibre vs. psyllium for chronic constipation. Aliment Pharmacol Ther. 2016 Jul;44(1):35-44. doi: 10.1111/apt.13647. Epub 2016 Apr 29. PMID 27125883
- [Result] Closa-Monasterolo R, Ferre N, Castillejo-DeVillasante G, Luque V, Gispert-Llaurado M, Zaragoza-Jordana M, Theis S, Escribano J. The use of inulin-type fructans improves stool consistency in constipated children. A randomised clinical trial: pilot study. Int J Food Sci Nutr. 2017 Aug;68(5):587-594. doi: 10.1080/09637486.2016.1263605. Epub 2016 Dec 8. PMID 27931142
- [Derived] Coss-Adame E, Garcia-Cedillo MF, Bustillo-Armendariz G, Huerta-de la Torre MF, Delgado-Bautista MK, Arenas-Martinez J, Cassis-Nosthas L. Agave tequilana Fructans Versus Psyllium plantago for Functional Constipation : Randomized Double-blind Clinical Trial. J Clin Gastroenterol. 2024 May-Jun 01;58(5):475-482. doi: 10.1097/MCG.0000000000001888. Epub 2023 Jul 3. PMID 37389917
- See also: Book — https://ciatej.mx/Sustainable-and-Integrated-Use-of-Agave.pdf
- See also: NOM-002-SAGARPA-2016 — http://vlex.com.mx/vid/relativa-caracteristicas-sanidad-calidad-655092789
- See also: Abstract — http://www.globalsciencebooks.info/Online/GSBOnline/images/0906/DBPBMB_3(SI1)/DBPBMB_3(SI1)59-64o.pdf
- See also: Article — http://pubs.acs.org/doi/abs/10.1021/jf060354v
- See also: Article — https://www.medigraphic.com/pdfs/medlab/myl-2009/myl099-10c.pdf
- See also: Article — https://www.researchgate.net/publication/259808612_Fructose_trehalose_and_sorbitol_malabsorption

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT04716868/Prot_SAP_000.pdf